CLINICAL TRIAL: NCT05471076
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Priming Regimens of 426c.Mod.Core-C4b and Optional Boost Regimen With HIV Trimer BG505 SOSIP.GT1.1 gp140, Both Adjuvanted With 3M-052-AF + Alum in Healthy, Adult Participants Without HIV
Brief Title: Trial to Evaluate the Safety and Immunogenicity of Priming Regimens of 426c.Mod.Core-C4b and Optional Boost Regimen With HIV Trimer BG505 SOSIP.GT1.1 gp140, Both Adjuvanted With 3M-052-AF + Alum in Healthy, Adult Participants Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 301
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Whether a participant receives a bolus dose or fractionated dose will be known, but randomization will occur within a given arm and both participants and clinicians will be blinded within a given arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Bolus Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose (Experimental): The Bolus Delivery Arm Group 1 will receive injections at 2 visits scheduled 3 months apart. At each injection visit the patient will get one dose divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Biological: 426c.Mod.Core-C4b 30 mcg; Biological: 426c.Mod.Core-C4b 100 mcg
- Bolus Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose (Experimental): The Bolus Delivery Arm Group 2 will receive injections at 2 visits scheduled 3 months apart. At each injection visit the patient will get one dose divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Biological: 426c.Mod.Core-C4b 100 mcg; Biological: 426c.Mod.Core-C4b 300 mcg
- Bolus Delivery, Group 3: First injection - Placebo, Final injection - Placebo (Placebo Comparator): The Bolus Delivery Arm Group 2 will receive injections at 2 visits scheduled 3 months apart. At each injection visit the patient will get one dose divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Other: Placebo
- Fractionated Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose (Experimental): The first dose for the Fractionated Delivery Arm Group 1 will be divided into 6 smaller amounts (2 visits per week for 3 weeks). The second dose will be given about 3 months later and will be given all at once. At each injection visit for the first dose, the patient will get one amount divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Biological: 426c.Mod.Core-C4b 30 mcg; Biological: 426c.Mod.Core-C4b 100 mcg
- Fractionated Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose (Experimental): The first dose for the Fractionated Delivery Arm Group 2 will be divided into 6 smaller amounts (2 visits per week for 3 weeks). The second dose will be given about 3 months later and will be given all at once. At each injection visit for the first dose, the patient will get one amount divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Biological: 426c.Mod.Core-C4b 100 mcg; Biological: 426c.Mod.Core-C4b 300 mcg
- Fractionated Delivery, Group 3: First injection - Placebo, Final injection - Placebo (Placebo Comparator): The first dose for the Fractionated Delivery Arm Group 2 will be divided into 6 smaller amounts (2 visits per week for 3 weeks). The second dose will be given about 3 months later and will be given all at once. At each injection visit for the first dose, the patient will get one amount divided into 2 injections - one in the deltoid muscle of each arm.
  Interventions: Other: Placebo
- Optional Boost Regimen with BG505 (Experimental): SOSIP.GT1.1 gp140
  Interventions: Biological: BG505

INTERVENTIONS:
Biological: 426c.Mod.Core-C4b 30 mcg — Administered via injection as a split dose into the deltoid muscle (both left and right).
  Other Names: Lower dose
  Arms: Bolus Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose; Fractionated Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose
Biological: 426c.Mod.Core-C4b 100 mcg — Administered via injection as a split dose into the deltoid muscle (both left and right).
  Other Names: Medium dose
  Arms: Bolus Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose; Bolus Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose; Fractionated Delivery, Group 1: First injection - Medium dose, Final injection - Lower dose; Fractionated Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose
Biological: 426c.Mod.Core-C4b 300 mcg — Administered via injection as a split dose into the deltoid muscle (both left and right).
  Other Names: Higher dose
  Arms: Bolus Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose; Fractionated Delivery, Group 2: First injection - Medium dose, Final injection - Higher dose
Other: Placebo — Administered via injection as a split dose into the deltoid muscle (both left and right).
  Arms: Bolus Delivery, Group 3: First injection - Placebo, Final injection - Placebo; Fractionated Delivery, Group 3: First injection - Placebo, Final injection - Placebo
Biological: BG505 — A soluble, cleavage-competent, trimeric HIV-1 envelope glycoprotein gp140 formulated at 2 mg/mL, 0.55 mL per vial, in 20 mM Tris, 100 mM NaCl, pH 7.5 will be admixed with 3M-052-AF (5 mcg) + Alum (500 mcg
  Arms: Optional Boost Regimen with BG505

SUMMARY:
The clinical study is designed to evaluate the ability of two priming vaccine regimens to activate and induce the maturation of cross-reactive CD4 binding site (CD4-bs) antibodies, including VRC01-class antibodies. VRC01- class antibodies are highly desirable to elicit via vaccination because they have broad cover all clades of HIV and passive administration of VRC01 monoclonal antibodies has been demonstrated to prevent acquisition of susceptible HIV strains in clinical trials. The study will assess whether B cells expressing VRC01-like B cell receptors proliferate following immunization with a 'germline-targeting' recombinant Env immunogen. The study will also test whether an immunization strategy based upon fractionated dose delivery of the immunogen may improve the maturation of VRC01-class B cells when compared to traditional bolus dosing. In addition, the study will test whether alterations in the dose of the subsequent boost immunizations affects VRC01-class B cell activation and the rate of antibody affinity maturation.

The primary hypothesis of the optional boost regimen is that BG505 SOSIP.GT1.1 gp140 adjuvated with 3M-052-AF + Alum is safe and well-tolerated and will further mature B-cell lineages elicited by 426c.Mod.Core-C4b priming regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of any questionnaire items answered incorrectly.
2. 18-55 years old, inclusive, on day of enrollment.
3. Available for clinic follow-up through the last clinic visit, willing to under go lymph node fine needle aspiration, and willing to be contacted 12 months after the last vaccine administration.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial.
5. In good general health according to the clinical judgement of the site investigator.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
7. Assessed as low risk for HIV acquisition per low risk guidelines, agrees to discuss HIV infection risks, agrees to risk reduction counseling, and agrees to avoid behavior associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed for 6 months or longer.
8. Hemoglobin:

   * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth
   * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months
   * ≥ 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months
   * For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth.
9. White blood cell (WBC) count > 3,500/mm3.
10. Platelets ≥125,000/mm3.
11. Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range.
12. Serum creatinine ≤1.1 x ULN based on the institutional normal range.
13. Blood pressure in the range of 90 to ≤ 150 mmHg systolic and 50 to ≤ 95 mmHg diastolic.
14. Negative results for HIV infection by an FDA-approved enzyme immunoassay(EIA) or chemiluminescent microparticle immunoassay (CMIA).
15. Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected.
16. Negative for Hepatitis B surface antigen.
17. For a volunteer capable of becoming pregnant:

    * Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their last vaccination timepoint.
    * Has negative β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment.

Exclusion Criteria:

1. Volunteer who is breast-feeding or pregnant.
2. Morbid Obesity. Enrollment of individuals with body mass index (BMI) ≥40, who the site investigator assesses are in good health, may be considered by PSRT on a case-by-case basis.
3. Diabetes mellitus (DM). Type 2 DM, controlled with diet alone, or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well-controlled on hypoglycemic agent(s) may be considered, provided the HgbA1c is ≤8% within the last 6 months (sites may draw these at screening).
4. International normalized ratio (INR) >1.2.
5. Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded).
6. Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions may be made by the PSRT for vaccines that have subsequently undergone licensure or Emergency Use Authorization by the FDA or, if outside the United States, by the national regulatory authority or World Health Organization. For volunteers who have received control/placebo in an experimental vaccine trial, the PSRT will determine eligibility on a case-by-case basis.
7. Systemic glucocorticoid use equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment, other systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, or congenital or acquired immunodeficiency.
8. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
9. Previous receipt of VRC01 monoclonal antibody.
10. Receipt of any live replicating vaccine within 4 weeks prior to enrollment. For receipt of ACAM2000 vaccine >28 days prior with a vaccination scab still present.
11. Receipt of any vaccines that are not covered in exclusion criterion #10 within 14 days prior to enrollment. Please note this includes replication incompetent vaccines such as the Jynneos vaccine for the prevention of monkeypox disease
12. Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
13. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
14. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any vaccine or any component of the study vaccine, including imidazoquinolone (eg, imiquimod).
15. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
16. Idiopathic urticaria within the past year.
17. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
18. Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
19. Asplenia or functional asplenia.
20. Active duty and reserve US military personnel.
21. Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, or cancer that, in the clinical judgement of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).
22. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]);
    * Uses more than one medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than one medication for maintenance therapy daily for greater than two years requires PSRT approval.
23. A participant with a history of an immune-mediated disease, either active or remote. Not exclusionary: 1) remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms, 2) mild psoriasis that does not require ongoing systemic treatment.
24. Investigator concern for difficulty with venous access based upon clinical history and physical examination. For example, history of IV drug abuse or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants showing local vaccination reactogenicity signs and symptoms | 14 days following each vaccination
  Assessed by clinic staff. For a given sign or symptom, each subject's reactogenicity will be counted once under the maximum severity for each injection/ vaccination.
Number of participants showing systemic vaccination reactogenicity signs and symptoms | 14 days following each vaccination
  Assessed by clinic staff. For a given sign or symptom, each subject's reactogenicity will be counted once under the maximum severity for each injection/ vaccination.
Number of serious adverse events (SAEs) | Through week 64
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of medically attended adverse events (MAAEs) | Through week 64
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of adverse events of special interest (AESIs) | Through week 64
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of AEs leading to early participant withdrawal or permanent discontinuation | Through week 64
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Frequency of CD4-bs-specific B cells | Through week 27
  Measured by flow cytometry analysis
Frequency of VRC01-like BCR sequences | Through week 27
  Determined by variable heavy chain domain (VH)/variable light chain domain (VL) sequencing of sorted B cells

SECONDARY OUTCOMES:
Response rate of Env-specific serum IgG binding antibodies. | Through week 27
Magnitude of Env-specific serum IgG binding antibodies. | Through week 27
Epitope-specificity of Env-specific serum IgG binding antibodies. | Through week 27
Avidity of Env-specific serum IgG binding antibodies. | Through week 27
Frequency of CD4-bs B cells and BCR sequences of isolated CD4-bs and VRC01-class memory B cells induced post-immunization with the traditional bolus dosing versus the fractionated dose delivery approach. | Through week 27
Frequency of CD4-bs B cells and BCR sequences of isolated CD4-bs and VRC01-class memory B cells induced post-immunization induced following a "low" or "high" dose second dose. | 14 days following second vaccination
Frequency of VRC01-class memory B cells induced post-immunization with the traditional bolus dosing versus the fractionated dose delivery approach. | Through week 27
Frequency of VRC01-class memory B cells induced following a "low" or "high" dose second dose. | 14 days following second vaccination
Response rate of serum antibody neutralization of the vaccine strain | 14 days following each vaccination
  Measured by TZM-bl assay.
Response rate of serum antibody neutralization of a panel of CD4-bs bnAb precursor-sensitive viruses. | 14 days following each vaccination
  Measured by TZM-bl assay.
Magnitude of serum antibody neutralization of the vaccine strain | 14 days following each vaccination
  Measured by TZM-bl assay.
Magnitude of serum antibody neutralization of a panel of CD4-bs bnAb precursor-sensitive viruses. | 14 days following each vaccination
  Measured by TZM-bl assay.
Comparison of CD4-bs-specific B cell frequencies in fractionated dosing versus traditional bolus dosing. | Through week 27
Comparison of BCR sequences frequencies in fractionated dosing versus traditional bolus dosing. | Through week 27
Response rate of VH/VL-pair sequence analysis of BCRs isolated from CD-4-bs-specific B cells | !4 days following each vaccination
Response rate of BG505 SOSIP.GT1.1 gp140 on the neutralizing activities of vaccine-induced antibodies in participants primed with 426c | Through week 27
Response rate of BG505 SOSIP.GT1.1 gp140 on the quality and quantity of Env-specific binding antibodies elicited after the GT1.1 immunization in participants primed with 426c | Through week 27
. Magnitude of BG505 SOSIP.GT1.1 gp140 on the quality and quantity of Env-specific binding antibodies elicited after the GT1.1 immunization in participants primed with 426c | Through week 27
Epitope specificity of BG505 SOSIP.GT1.1 gp140 on the quality and quantity of Env-specific binding antibodies elicited after the GT1.1 immunization in participants primed with 426c | Through week 27
Comparison of CD4-bs antibodies isolated after the GT.1 immunization, as compared to those elicited by the 426c | Through week 27
Response rate of BG505 SOSIP.GT1.1 gp140 on the CD4+ T cell response in participants primed with 426c | Through week 27
Magnitude of BG505 SOSIP.GT1.1 gp140 on the CD4+ T cell response in participants primed with 426c | Through week 27

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Scott, MD, Study Chair — University of California, San Francisco; Kristen Cohen, MD, Study Chair — Fred Hutch Cancer Center, Seattle, WA
Locations (6):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Libera M, Caputo V, Laterza G, Moudoud L, Soggiu A, Bonizzi L, Diotti RA. The Question of HIV Vaccine: Why Is a Solution Not Yet Available? J Immunol Res. 2024 Apr 8;2024:2147912. doi: 10.1155/2024/2147912. eCollection 2024. PMID 38628675